CLINICAL TRIAL: NCT06766864
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study Evaluating the Safety and Pharmacokinetics of Subcutaneous Administration of Single Ascending Doses of DR-01 in Healthy Volunteers
Brief Title: A Study of Subcutaneous DR-01 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dren Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR-01-HV-001
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- DL1 of DR-01 (Experimental): Subjects in this arm will receive a single dose of dose level 1 of DR-01
  Interventions: Drug: DR-01
- DL2 of DR-01 (Experimental): Subjects in this arm will receive a single dose of dose level 2 of DR-01
  Interventions: Drug: DR-01
- DL3 of DR-01 (Experimental): Subjects in this arm will receive a single dose of dose level 3 of DR-01
  Interventions: Drug: DR-01
- Placebo (Placebo Comparator): Subjects in this arm will receive a single dose of placebo
  Interventions: Other: Placebo
- DL4 of DR-01 (Experimental): Subjects in this arm will receive a single dose of dose level 4 of DR-01
  Interventions: Drug: DR-01

INTERVENTIONS:
Drug: DR-01 — DR-01 is a monoclonal antibody
  Arms: DL1 of DR-01; DL2 of DR-01; DL3 of DR-01; DL4 of DR-01
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, Phase 1 study to evaluate the safety, tolerability, PK, immunogenicity, and PD of SC administration of single ascending doses of DR-01 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, in the opinion of the Investigator, as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead ECGs. A subject with a clinical abnormality or laboratory parameter(s) outside the reference range that is not specifically listed in the inclusion or exclusion criteria may be included if the Investigator (in consultation with the Medical Monitor) agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures, subject safety, or data interpretation.
2. Between 18 and 65 years of age, inclusive, of any race or gender.
3. Body weight at screening ≥ 40 kg and < 120 kg, with body mass index between 18 and 35 kg/m2.
4. Adequate abdominal adipose tissue for SC injection.
5. Ability to understand and comply with protocol-required study procedures, including admission to the Clinical Research Unit the day prior to dosing with an overnight stay, and voluntarily sign a written informed consent document.
6. Use of a highly effective contraceptive measure (< 1% failure rate; see Section 13.1) for all males and all females of childbearing potential during study and 90 days postdose for males and 30 days postdose for females. Bilateral tubal ligation performed 6 months prior to screening is considered a highly effective contraceptive measure for female subjects and female partners of male subjects and does not require the use of additional contraception. Females of childbearing potential must have a confirmatory negative urine pregnancy test on Day -1/prior to dosing on Day 1. Females who are not of childbearing potential (i.e., who are considered to be postmenopausal [≥ 12 months of non-therapy amenorrhea] or surgically sterile [absence of ovaries and/or uterus or bilateral tubal ligation]) are not required to have a pregnancy test or use contraception.

Exclusion Criteria:

1. History or presence of a disease or condition that, in the Investigator's opinion, constitutes a risk when taking study drug or interfering with study assessment or interpretation of the data.
2. Medical history of severe allergic reaction, angioedema, anaphylaxis, clinically significant drug hypersensitivity reaction, or autoimmune or immunodeficiency disorder.
3. History of malignant neoplasm within 5 years prior to screening, except for fully treated nonmetastatic basal or squamous cell cancers of the skin (within 3 years) that shows no evidence of recurrence.
4. Any of the following types of infection within 28 days of screening or before randomization:

   1. Serious (requiring hospitalization, and/or IV antimicrobial treatment).
   2. Chronic (duration of symptoms, signs, and/or treatment of 6 weeks or longer).
   3. Viral reactivation of CMV, EBV, VZV, or HSV type infection requiring systemic therapy in the last 2 years. Periodic HSV viral reactivation (e.g., cold sore) treated with a short course of systemic antiviral therapy within the last 2 years would not be exclusionary.
5. Any of the following:

   1. HIV.
   2. Current infection with HBV (i.e., positive for HBsAg and/or polymerase chain reaction positive for HBV DNA).
   3. Current infection with HCV (i.e., positive for HCV RNA).
   4. Active infection with SARS-CoV-2.
6. Untreated latent tuberculosis infection, as indicated by IFNγ release assay, without documentation of appropriate treatment (as defined by the World Health Organization and/or the US Centers for Disease Control and Prevention).
7. Any surgical procedure (except for minor surgery requiring local or no anesthesia and without any complications or sequelae) within 12 weeks prior to screening or any planned surgical procedure during the study.
8. Use of prescription or non-prescription drugs (including recreational drugs, herbal medications, vitamins, and supplements) within 7 days or 5 half-lives (whichever is longer) prior to dosing, unless in the opinion of the Investigator (in consultation with the Medical Monitor), the medication will not interfere with the study or compromise subject safety. Paracetamol (acetaminophen) at doses of ≤ 4 grams/day, and occasional use of non-steroidal anti-inflammatory drugs at labeled/approved doses, are permitted.
9. Live or live-attenuated vaccination within 28 days prior to dosing on Day 1 or during the study. All non-live vaccines (e.g., flu or COVID-19) are permitted.
10. Previous exposure to DR-01.
11. Known hypersensitivity to biologics.
12. Prior anaphylaxis to a biological agent or vaccine.
13. Neutrophil or lymphocyte counts below the normal range at screening; subjects who meet this exclusion criterion will be allowed to retest during screening, with at least a 1-week interval between the date of the first failed test and the date of the subsequent test.
14. Estimated glomerular filtration rate by Chronic Kidney Disease Epidemiology Collaboration equation calculation ≤ 60 mL/min/1.73 m2 at screening, provided no signs of kidney damage such as proteinuria; subjects who meet this exclusion criterion will be allowed to retest during screening, with at least a 1-week interval between the date of the first failed test and the date of the subsequent test.
15. Alanine transaminase and/or aspartate aminotransferase > 2 × ULN and total bilirubin > 1.5 × ULN (> 3 × ULN if known Gilbert's disease) at screening; subjects who meet this exclusion criterion will be allowed to retest during screening, with at least a 1-week interval between the date of the first failed test and the date of the subsequent test.
16. Other clinically significant abnormalities of laboratory assessments, as judged by the Investigator and/or Medical Monitor, that could affect the safety of the subject, or the interpretation of study data.
17. ECG QTcF > 490 msec.
18. Participation in a clinical trial and has received an investigational product within the following time period prior to screening in the current study: 3 months (for biologic therapies) or 1 month (for non-biologic therapies), 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
19. Exposure to more than 4 new chemical entities within 12 months prior to dosing on Day 1.
20. Participation in a clinical trial resulting in loss of blood or blood products in excess of 500 mL within 3 months prior to screening.
21. Women who are currently pregnant or breastfeeding, or who intend to become pregnant or to breastfeed at any time during the study or within 30 days postdose.
22. Positive drug screen at screening or on Day -1/prior to dosing on Day 1, with the exception of a positive result for THC, as recreational use of cannabis is allowed.
23. Positive alcohol screen on Day -1/prior to dosing on Day 1; females are allowed up to 7 units of alcohol per week and males are allowed up to 14 units of alcohol per week after collection of the 24-hour post-dose PK sample.
24. Unstable lifestyle factors (including but not limited to excessive alcohol use, heavy nicotine use [cigarettes or vaping; heavy use is defined as ≥ 1 pack of cigarettes/day], or substance abuse) that, in the opinion of the Investigator, would interfere with the ability of a subject to complete the study.
25. Any other medical or psychiatric condition, or laboratory abnormality that would, in the opinion of the Investigator or Medical Monitor, increase the subject's risk of participation, jeopardize completion of the study, or compromise interpretation of the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events [Safety and Tolerability] as assessed by CTCAE v5.0 after a single SC dose | Up to 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rothenberg, MD, PhD, Study Director — Dren Bio
Locations (1):
- Dren Investigational Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No